CLINICAL TRIAL: NCT06518980
Title: Prospective Validation of Intraoperative Blood Pressure Monitors: the Influence of Site and Execution Strategy. The PROMISES Trial
Brief Title: Prospective Validation of Intraoperative Blood Pressure Monitors
Acronym: PROMISES
Status: Not yet recruiting | Type: Observational
Sponsor: Ciusss de L'Est de l'Île de Montréal (Other)
Responsible Party: Principal Investigator, Pascal Laferrière-Langlois, MD, MSc, FRQS, Assistant Professor, Principal Investigator, Anesthesiologist, Ciusss de L'Est de l'Île de Montréal
Other Study IDs: 2025-3776
Record Dates: First submitted 2024-07-09; First posted 2024-07-25 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Anesthesia; Blood Pressure
Keywords: anesthesia; blood pressure; noninvasive blood pressure; invasive blood pressure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This observational study aims to identify the incidence and importance of discrepancies between measurements of intraoperative invasive and noninvasive blood pressure monitoring in patients undergoing non-cardiac surgeries under general anesthesia . The main questions it aims to answer are :

* The importance of the differences, in mmHg, between the non-invasive and invasive blood pressure measurements (NIBP-IBP) on systolic, diastolic and mean arterial pressure.
* Identify the predictive factors associated with these differences.

DETAILED DESCRIPTION:
The monitoring of arterial blood pressure, invasively or noninvasively, is a requirement for perioperative hemodynamic and anesthesia management to optimize the administration of fluids and vasopressors. Numerous trials have highlighted the consequences of intraoperative blood pressure variability regarding the risk of serious complications and postoperative mortality associated with organ ischemia, and bleeding. Precisely, intraoperative hypotension (MAP <65 mm Hg) has been associated with cardiac complications as well as acute kidney injury. While no optimal intraoperative blood pressure targets has been established to minimize perioperative complications, a recent comprehensive literature review established recommended mean arterial pressure (MAP), and blood pressure (BP) targets within 100% to 120% of BP baseline with MAP ≥60 mm Hg if the patient presented low baseline (systolic BP <90 mm Hg or diastolic BP <50 mm Hg), and MAP within 90% to 110% BP baseline and ≈65 to 95 mm Hg for normal baseline (systolic BP 90-129 mm Hg and diastolic BP 50-79 mm Hg) patients.

Invasive blood pressure monitoring by arterial catheterization is the gold standard in intraoperative hemodynamic management. While providing continuous blood pressure readings allowing for dynamic and constant monitoring, clinically relevant transducer inaccuracies have been documented, present in up to 30% of patients. Within patients of the same study, comparison of invasive and noninvasive blood pressure demonstrated considerable overestimation of systolic blood pressure and underestimation of diastolic blood pressure.

Oscillometric blood pressure monitoring is noninvasive, quick, and effortless.Despite its convenience, the oscillometric monitoring of blood pressure does not allow for continuous blood pressure measurement, possibly delaying or missing the recognition of hypotensive episodes. Moreover, oscillometric devices can tend to inaccurately measure blood pressure in comparison to invasive monitoring methods. In intraoperative and critical care settings, studies have shown oscillometric devices' tendencies to overestimate low blood pressure, failing to accurately detect hypotensive episodes, thus demonstrating the superiority of invasive monitoring methods.

The discrepancies between invasive and noninvasive methods of blood pressure monitoring have been described in prior studies. It has been determined that noninvasive blood pressure tended to be greater than invasive blood pressure in 56.1% of systolic measurements, and 67.3% of diastolic measurements for the same patient. Furthermore, noninvasive blood pressure readings tend to overestimate mean arterial pressure for low blood pressure values, and to underestimate mean arterial pressure for high blood pressure values.

Considering the consequences associated with even short intraoperative hypotensive episodes, the discrepancies between noninvasive and invasive blood pressure monitoring are not negligible. Currently, little is known about the relation between these discrepancies and contextual elements linked to the patient or the surgery.

Therefore, this prospective observational trial aims to identify the incidence of gradients between intraoperative noninvasive and invasive blood pressure monitoring and extract key relationships between the occurrence of these gradients and the patient's comorbidity profile, the monitor's parameters and artifacts, and the perioperative chronology.

Study duration: 12 months

Study Center: Maisonneuve-Rosemont Hospital, Integrated University Health and Social Services Centre (CIUSSS) de l'Est de l'Ile de Montreal (CEMTL), University of Montreal, Montreal, Quebec, Canada.

Adverse Events: there is very little risk involved with participation in this study, side effects that may be associated with the use of intra-radial canula for invasive blood pressure measurement.

ELIGIBILITY:
Inclusion Criteria:

* Fully consented, adult patients above 18 years old;
* Undergoing surgery of duration time expected at least 60 minutes using general anesthesia;
* Supine positioning during the surgery;
* Surgery requiring an arterial line;
* Both arms available for instrumentation during the surgery.

Exclusion Criteria:

* Atrial fibrillation, multifocal atrial tachycardia, or any other irregular hear rythm;
* Gradient of mean arterial pressure between the two arms greater than 5 mm Hg, as measured during the recruitment process.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing non-cardiac elective surgery expected to last at least 60 minutes, under general anesthesia, and to require an arterial line.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Difference between non-invasive blood pressure (NIBP) and invasive blood pressure (IBP) measurements | Time Frame: from arrival in preoperative unit patient's departure from PACU and/or removal of IBP device, expected duration approximately between 2 and 8 hours
  Describe the difference, in mm of Hg, between intraoperative monitoring of noninvasive and invasive blood (NIBP-IBP) on systolic, diastolic and mean arterial pressures
Predictive factors associated with the between non-invasive blood pressure (NIBP) and invasive blood pressure (IBP) measurement differences | Time Frame: From patient file analysis at time of recruitment until patient's departure from PACU and/or removal of IBP device, expected duration approximately a year.
  Identify predictive factors (such as patient, surgery, and anesthesia characteristics) statistically associated with the appearance of NIBP-IBP measurement differences

SECONDARY OUTCOMES:
Comparison of preoperative NIBP and pre-induction NIBP | From installation of non-invasive blood pressure (NIBP) device in preop until installation of arterial line, pre-induction. Expected duration approximately between 1 and 2 hours.
  Compare preoperative non-invasive blood pressure (NIBP) measurements prior to the surgery and the average pre-induction NIBP recorded in the operating room
Compare the discrepancies between non-invasive blood pressure (NIBP) and invasive blood pressure (IBP) measurements to the accuracy standards of the Association for the Advancement of Medical Instrumentation | From installation of patient's arterial line until removal of patient's arterial line, expected duration approximately between 1 and 8 hours.
  Compare the NIBP-IBP discrepancy to the accuracy standards of the Association for the Advancement of Medical Instrumentation (AAMI): a maximal mean difference of 5 mm Hg and a standard deviation of 8 mm Hg.
Impact of patient comorbidities (age, weight, height, BMI, heart condition, vascular condition) on occurrences of discrepancies between non-invasive blood pressure (NIBP) and invasive blood pressure (IBP) measurements | From patient file analysis at time of recruitment until the end of statistical analysis. Expected duration: up to a year.
  Evaluate the impact of patient's characteristics and comorbidities collected via REDCap questionnaire (age, weight, height, BMI, heart condition, vascular condition) on the occurrence of NIBP-IBP discrepancies.
Statistical correlation between radial artery ultrasound measurements on the occurrence of discrepancies between non-invasive blood pressure (NIBP) and invasive blood pressure (IBP) measurements | From measurement of patient's radial artery via ultrasonography before induction until the end of statistical analysis. Expected duration: up to a year.
  Evaluate the impact, via statistical analysis, of radial artery ultrasound characteristics (inter-intima diameter, velocity) on the occurrence of NIBP-IBP discrepancies.
Statistical correlation between administration of vasoactive drugs and fluids on the occurrence of discrepancies between non-invasive blood pressure (NIBP) and invasive blood pressure (IBP) measurements | From administration of first fluid or vasoactive drug until patient's departure from PACU and/or removal of arterial line. Expected duration between 2 and 8 hours.
  Evaluate the impact, via statistical analysis, of vasoactive drug administration and fluid (phenylephrine, ephedrine) administration on the occurrence of NIBP-IBP discrepancies
Statistical correlation between surgical characteristics (approach, duration, type of surgery, etc) on the occurrence of discrepancies between non-invasive blood pressure (NIBP) and invasive blood pressure (IBP) measurements | From patient file analysis at time of recruitment until the end of statistical analysis. Expected duration up to a year.
  Evaluate the impact, via statistical analysis, of surgical characteristics (approach, duration, type of surgery, etc) on the occurrence of NIBP-IBP measurement discrepancies.
Statistical correlation between anesthesia condition on the occurrence of discrepancies between non-invasive blood pressure (NIBP) and invasive blood pressure (IBP) measurements | From anesthesia induction until patient's departure from PACU and/or removal of arterial line, expected duration between 2 and 8 hours.
  Evaluate the impact of anesthesia condition (depth of anesthesia, nociception level) on the occurrence of NIBP-IBP discrepancies.
Describe the incidence of overdamping and underdamping upon installation of the arterial line | from installation of radial line until removal of arterial line. Expected duration between 5 and 15 minutes.
  Describe the incidence of overdamping and underdamping upon installation of the arterial line
Describe the impact of overdamping and underdamping upon installation of the arterial line on the occurrence of discrepancies between non-invasive blood pressure (NIBP) and invasive blood pressure (IBP) measurements | Time Frame : from installation of radial line until removal of radial line. Expected duration between 1 and 8 hours.
  Describe the impact of overdamping and underdamping upon installation of the arterial line on the occurrence of NIBP-IBP discrepancies
Evaluate statistical correlation between anesthesiologist's confidence in the arterial line, and importance of discrepancies between non-invasive blood pressure (NIBP) and invasive blood pressure (IBP) measurements | from installation of radial line until patient's departure from PACU and/or removal of arterial line. Expected duration between 1 andd 8 hours.
  Evaluate the relation between the healthcare provider's confidence in the arterial line and the presence and importance of NIBP-IBP discrepancies. Confidence will be assessed at 30 minute intervals during the surgery by offering multiple choices for confidence ranking. Confidence scale will be as follows: 0= no trust in radial line, 1= weak trust in radial line, 2= moderate trust in radial line, 3=strong trust in radial line, 4= absolute trust in radial line

CONTACTS AND LOCATIONS:
Overall Officials: Pascal Laferrière-Langlois, Principal Investigator — Ciusss de L'Est de l'Île de Montréal
Locations (1):
- Maisonneuve-Rosemont Hospital - CIUSSS de l'Est de l'Île de Montréal, Montreal East, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Meng L, Yu W, Wang T, Zhang L, Heerdt PM, Gelb AW. Blood Pressure Targets in Perioperative Care. Hypertension. 2018 Oct;72(4):806-817. doi: 10.1161/HYPERTENSIONAHA.118.11688. No abstract available. PMID 30354725
- [Background] Mascha EJ, Yang D, Weiss S, Sessler DI. Intraoperative Mean Arterial Pressure Variability and 30-day Mortality in Patients Having Noncardiac Surgery. Anesthesiology. 2015 Jul;123(1):79-91. doi: 10.1097/ALN.0000000000000686. PMID 25929547
- [Background] Tassoudis V, Vretzakis G, Petsiti A, Stamatiou G, Bouzia K, Melekos M, Tzovaras G. Impact of intraoperative hypotension on hospital stay in major abdominal surgery. J Anesth. 2011 Aug;25(4):492-9. doi: 10.1007/s00540-011-1152-1. Epub 2011 May 6. PMID 21547554
- [Background] Salmasi V, Maheshwari K, Yang D, Mascha EJ, Singh A, Sessler DI, Kurz A. Relationship between Intraoperative Hypotension, Defined by Either Reduction from Baseline or Absolute Thresholds, and Acute Kidney and Myocardial Injury after Noncardiac Surgery: A Retrospective Cohort Analysis. Anesthesiology. 2017 Jan;126(1):47-65. doi: 10.1097/ALN.0000000000001432. PMID 27792044
- [Background] Sun LY, Wijeysundera DN, Tait GA, Beattie WS. Association of intraoperative hypotension with acute kidney injury after elective noncardiac surgery. Anesthesiology. 2015 Sep;123(3):515-23. doi: 10.1097/ALN.0000000000000765. PMID 26181335
- [Background] Walsh M, Devereaux PJ, Garg AX, Kurz A, Turan A, Rodseth RN, Cywinski J, Thabane L, Sessler DI. Relationship between intraoperative mean arterial pressure and clinical outcomes after noncardiac surgery: toward an empirical definition of hypotension. Anesthesiology. 2013 Sep;119(3):507-15. doi: 10.1097/ALN.0b013e3182a10e26. PMID 23835589
- [Background] van Waes JA, van Klei WA, Wijeysundera DN, van Wolfswinkel L, Lindsay TF, Beattie WS. Association between Intraoperative Hypotension and Myocardial Injury after Vascular Surgery. Anesthesiology. 2016 Jan;124(1):35-44. doi: 10.1097/ALN.0000000000000922. PMID 26540148
- [Background] Botto F, Alonso-Coello P, Chan MT, Villar JC, Xavier D, Srinathan S, Guyatt G, Cruz P, Graham M, Wang CY, Berwanger O, Pearse RM, Biccard BM, Abraham V, Malaga G, Hillis GS, Rodseth RN, Cook D, Polanczyk CA, Szczeklik W, Sessler DI, Sheth T, Ackland GL, Leuwer M, Garg AX, Lemanach Y, Pettit S, Heels-Ansdell D, Luratibuse G, Walsh M, Sapsford R, Schunemann HJ, Kurz A, Thomas S, Mrkobrada M, Thabane L, Gerstein H, Paniagua P, Nagele P, Raina P, Yusuf S, Devereaux PJ, Devereaux PJ, Sessler DI, Walsh M, Guyatt G, McQueen MJ, Bhandari M, Cook D, Bosch J, Buckley N, Yusuf S, Chow CK, Hillis GS, Halliwell R, Li S, Lee VW, Mooney J, Polanczyk CA, Furtado MV, Berwanger O, Suzumura E, Santucci E, Leite K, Santo JA, Jardim CA, Cavalcanti AB, Guimaraes HP, Jacka MJ, Graham M, McAlister F, McMurtry S, Townsend D, Pannu N, Bagshaw S, Bessissow A, Bhandari M, Duceppe E, Eikelboom J, Ganame J, Hankinson J, Hill S, Jolly S, Lamy A, Ling E, Magloire P, Pare G, Reddy D, Szalay D, Tittley J, Weitz J, Whitlock R, Darvish-Kazim S, Debeer J, Kavsak P, Kearon C, Mizera R, O'Donnell M, McQueen M, Pinthus J, Ribas S, Simunovic M, Tandon V, Vanhelder T, Winemaker M, Gerstein H, McDonald S, O'Bryne P, Patel A, Paul J, Punthakee Z, Raymer K, Salehian O, Spencer F, Walter S, Worster A, Adili A, Clase C, Cook D, Crowther M, Douketis J, Gangji A, Jackson P, Lim W, Lovrics P, Mazzadi S, Orovan W, Rudkowski J, Soth M, Tiboni M, Acedillo R, Garg A, Hildebrand A, Lam N, Macneil D, Mrkobrada M, Roshanov PS, Srinathan SK, Ramsey C, John PS, Thorlacius L, Siddiqui FS, Grocott HP, McKay A, Lee TW, Amadeo R, Funk D, McDonald H, Zacharias J, Villar JC, Cortes OL, Chaparro MS, Vasquez S, Castaneda A, Ferreira S, Coriat P, Monneret D, Goarin JP, Esteve CI, Royer C, Daas G, Chan MT, Choi GY, Gin T, Lit LC, Xavier D, Sigamani A, Faruqui A, Dhanpal R, Almeida S, Cherian J, Furruqh S, Abraham V, Afzal L, George P, Mala S, Schunemann H, Muti P, Vizza E, Wang CY, Ong GS, Mansor M, Tan AS, Shariffuddin II, Vasanthan V, Hashim NH, Undok AW, Ki U, Lai HY, Ahmad WA, Razack AH, Malaga G, Valderrama-Victoria V, Loza-Herrera JD, De Los Angeles Lazo M, Rotta-Rotta A, Szczeklik W, Sokolowska B, Musial J, Gorka J, Iwaszczuk P, Kozka M, Chwala M, Raczek M, Mrowiecki T, Kaczmarek B, Biccard B, Cassimjee H, Gopalan D, Kisten T, Mugabi A, Naidoo P, Naidoo R, Rodseth R, Skinner D, Torborg A, Paniagua P, Urrutia G, Maestre ML, Santalo M, Gonzalez R, Font A, Martinez C, Pelaez X, De Antonio M, Villamor JM, Garcia JA, Ferre MJ, Popova E, Alonso-Coello P, Garutti I, Cruz P, Fernandez C, Palencia M, Diaz S, Del Castillo T, Varela A, de Miguel A, Munoz M, Pineiro P, Cusati G, Del Barrio M, Membrillo MJ, Orozco D, Reyes F, Sapsford RJ, Barth J, Scott J, Hall A, Howell S, Lobley M, Woods J, Howard S, Fletcher J, Dewhirst N, Williams C, Rushton A, Welters I, Leuwer M, Pearse R, Ackland G, Khan A, Niebrzegowska E, Benton S, Wragg A, Archbold A, Smith A, McAlees E, Ramballi C, Macdonald N, Januszewska M, Stephens R, Reyes A, Paredes LG, Sultan P, Cain D, Whittle J, Del Arroyo AG, Sessler DI, Kurz A, Sun Z, Finnegan PS, Egan C, Honar H, Shahinyan A, Panjasawatwong K, Fu AY, Wang S, Reineks E, Nagele P, Blood J, Kalin M, Gibson D, Wildes T; Vascular events In noncardiac Surgery patIents cOhort evaluatioN (VISION) Writing Group, on behalf of The Vascular events In noncardiac Surgery patIents cOhort evaluatioN (VISION) Investigators; Appendix 1. The Vascular events In noncardiac Surgery patIents cOhort evaluatioN (VISION) Study Investigators Writing Group; Appendix 2. The Vascular events In noncardiac Surgery patIents cOhort evaluatioN Operations Committee; Vascular events In noncardiac Surgery patIents cOhort evaluatioN VISION Study Investigators. Myocardial injury after noncardiac surgery: a large, international, prospective cohort study establishing diagnostic criteria, characteristics, predictors, and 30-day outcomes. Anesthesiology. 2014 Mar;120(3):564-78. doi: 10.1097/ALN.0000000000000113. PMID 24534856
- [Background] Wijnberge M, Schenk J, Bulle E, Vlaar AP, Maheshwari K, Hollmann MW, Binnekade JM, Geerts BF, Veelo DP. Association of intraoperative hypotension with postoperative morbidity and mortality: systematic review and meta-analysis. BJS Open. 2021 Jan 8;5(1):zraa018. doi: 10.1093/bjsopen/zraa018. PMID 33609377
- [Background] Roach JK, Thiele RH. Perioperative blood pressure monitoring. Best Pract Res Clin Anaesthesiol. 2019 Jun;33(2):127-138. doi: 10.1016/j.bpa.2019.05.001. Epub 2019 May 7. PMID 31582093
- [Background] Romagnoli S, Ricci Z, Quattrone D, Tofani L, Tujjar O, Villa G, Romano SM, De Gaudio AR. Accuracy of invasive arterial pressure monitoring in cardiovascular patients: an observational study. Crit Care. 2014 Nov 30;18(6):644. doi: 10.1186/s13054-014-0644-4. PMID 25433536
- [Background] Truijen J, van Lieshout JJ, Wesselink WA, Westerhof BE. Noninvasive continuous hemodynamic monitoring. J Clin Monit Comput. 2012 Aug;26(4):267-78. doi: 10.1007/s10877-012-9375-8. Epub 2012 Jun 14. PMID 22695821
- [Background] Naylor AJ, Sessler DI, Maheshwari K, Khanna AK, Yang D, Mascha EJ, Suleiman I, Reville EM, Cote D, Hutcherson MT, Nguyen BM, Elsharkawy H, Kurz A. Arterial Catheters for Early Detection and Treatment of Hypotension During Major Noncardiac Surgery: A Randomized Trial. Anesth Analg. 2020 Nov;131(5):1540-1550. doi: 10.1213/ANE.0000000000004370. PMID 33079877
- [Background] Wax DB, Lin HM, Leibowitz AB. Invasive and concomitant noninvasive intraoperative blood pressure monitoring: observed differences in measurements and associated therapeutic interventions. Anesthesiology. 2011 Nov;115(5):973-8. doi: 10.1097/ALN.0b013e3182330286. PMID 21952254
- [Background] Meidert AS, Dolch ME, Muhlbauer K, Zwissler B, Klein M, Briegel J, Czerner S. Oscillometric versus invasive blood pressure measurement in patients with shock: a prospective observational study in the emergency department. J Clin Monit Comput. 2021 Apr;35(2):387-393. doi: 10.1007/s10877-020-00482-2. Epub 2020 Feb 13. PMID 32056094
- [Background] Rutten AJ, Ilsley AH, Skowronski GA, Runciman WB. A comparative study of the measurement of mean arterial blood pressure using automatic oscillometers, arterial cannulation and auscultation. Anaesth Intensive Care. 1986 Feb;14(1):58-65. doi: 10.1177/0310057X8601400113. PMID 3954015
- [Background] Gabriel A, Lindblad LE, Angleryd C. Non-invasive vs. invasive beat-to-beat monitoring of blood pressure. Clin Physiol. 1992 Mar;12(2):229-35. doi: 10.1111/j.1475-097x.1992.tb00309.x. PMID 1582140
- [Background] Francke A, Wachsmuth H. [How accurate is invasive blood pressure determination with fluid-filled pressure line systems?]. Anaesthesiol Reanim. 2000;25(2):46-54. German. PMID 10816897
- [Background] Mireles SA, Jaffe RA, Drover DR, Brock-Utne JG. A poor correlation exists between oscillometric and radial arterial blood pressure as measured by the Philips MP90 monitor. J Clin Monit Comput. 2009 Jun;23(3):169-74. doi: 10.1007/s10877-009-9178-8. Epub 2009 Apr 25. PMID 19396553
- [Background] Ribezzo S, Spina E, Di Bartolomeo S, Sanson G. Noninvasive techniques for blood pressure measurement are not a reliable alternative to direct measurement: a randomized crossover trial in ICU. ScientificWorldJournal. 2014 Jan 30;2014:353628. doi: 10.1155/2014/353628. eCollection 2014. PMID 24616624
- [Background] Velasco A, Ono C, Nugent K, Tarwater P, Kumar A. Ultrasonic evaluation of the radial artery diameter in a local population from Texas. J Invasive Cardiol. 2012 Jul;24(7):339-41. PMID 22781473
- [Background] Pancholy SB, Shah S, Patel TM. Radial Artery Access, Hemostasis, and Radial Artery Occlusion. Interv Cardiol Clin. 2015 Apr;4(2):121-125. doi: 10.1016/j.iccl.2015.01.004. Epub 2015 Mar 31. PMID 28582044
- See also: Guidelines to Anesthesia | Canadian Anesthesiologists' Society. — http://cas.ca/en/practice-resources/guidelines-to-anesthesia
- See also: Coronary Interventions Handbook ; An Interventional Council Review — https://www.acc.org/membership/features/coronary-interventions-handbook
- See also: Bickley, Lynn S. Bates' Guide to Physical Examination and History Taking. Philadelphia: Lippincott Williams & Wilkins, 2020. — https://shop.lww.com/Bates--Guide-To-Physical-Examination-and-History-Taking-13e-with-Videos-Lippincott-Connect-Print-Book-and-Digi/p/9781975210878
- See also: 26. Schroeder, Becky, et al. "Chapter 36 - Cardiovascular Monitoring." Miller's Anesthesia, Elsevier, Philadelphia, Pennsylvania , 2020, pp. 1145-1193. From Gropper, Michael A., and Ronald D. Miller. Miller's Anesthesia. Elsevier, 2020. — https://shop.elsevier.com/books/millers-anesthesia-2-volume-set/gropper/978-0-323-59604-6